CLINICAL TRIAL: NCT00953771
Title: Phase II Study of Danazol With Plasma Exchange and Steroids for the Treatment of Thrombotic Thrombocytopenic Purpura
Brief Title: Safety Study of Danazol With Plasma Exchange and Steroids for the Treatment of Thrombotic Thrombocytopenic Purpura (TTP)
Acronym: TTP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Beth Israel Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Shapira, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2608; 055-08 (Other: Beth Israel Medical Center)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2023-08-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: TTP; Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Danazol; Plasma Exchange; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Danazol, Plex, Steroids (Experimental): Everyone will receive Danazol with plasma exchange and corticosteroids
  Interventions: Drug: Danazol
- Historic Control (No Intervention)

INTERVENTIONS:
Drug: Danazol — Danazol 600 mg PO will be initiated with plasma exchange and corticosteroids at the time of enrollment.
  Other Names: Plasma Exchange; Corticosteroids
  Arms: Danazol, Plex, Steroids

SUMMARY:
The purpose of the study is to find out if administration of danazol with plasma exchange and corticosteroids will reduce the number of plasma exchanges required to control Thrombotic Thrombocytopenic Purpura (TTP).

DETAILED DESCRIPTION:
Danazol is a synthetic steroid hormone structurally resembling a group of natural hormones (androgens)found in the body. Danazol has immune modifying activity and is effective in treatment of blood disorders with low platelet counts such as idiopathic thrombocytopenic purpura (however FDA has not yet approved danazol for this disorder). A study of danazol in conjunction with plasma exchange for thrombotic thrombocytopenic purpura showed that danazol decreased the number of plasma exchanges required by approximately 80% and reduced the time needed to control the disease. It's not clear how danazol works in TTP. It is not approved by the FDA for the treatment of TTP.

ELIGIBILITY:
Inclusion Criteria:

* TTP with platelets less than 100,000 and microangiopathic hemolytic anemia
* Age greater than 18 and less than 60
* LDH > 2x upper limit of normal
* PT and PTT normal
* Patients must give signed informed consent
* Pre-menopausal woman must have negative pregnancy test.
* TTP not related to underlying cancer, treatment of cancer or transplantation.
* TTP not associated with drugs.

Exclusion Criteria:

* LFTs AST/ALT > 2x upper limit of normal
* Hepatitis B and Hepatitis C infection.
* HIV with active opportunistic infections
* Acute or chronic Disseminated Intravascular Coagulation (DIC), defined as D-dimer 8ug/ml and fibrinogen<100 mg/dl
* TTP related to drugs, malignancy and transplantation.
* Pregnancy
* Concurrent other investigational drug use during this study.
* Porphyria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2015-11-19 (Actual); Study Completion 2015-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Shapira, M.D., Principal Investigator — Mount Sinai St. Luke's-Roosevelt
Locations (1):
- Mount Sinai St. Luke's-Roosevelt, New York, New York, United States

REFERENCES:
- [Result] Torri V, Friedman M, Shapira I, Patel AA, Yoe J, Shah VP, Mirzoyev T, Machuca M, Varma M. Phase II study of danazol with plasma exchange and corticosteroids for the treatment of thrombotic thrombocytopenic purpura. Blood (2023) 142 (Supplement 1): 4007.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened for patient recruitment on Oct 29, 2008 at Beth Israel Medical Center and St. Luke's-Roosevelt Hospital Center. The study was closed by the IRB on 10/12/2018 due to low enrollment. The last date of study data collection was 11/19/2015.
Pre-assignment Details: Subjects were not enrolled to the control group; data was retrospectively collected by viewing the charts of 20 patients who received Plasma Exchange
Groups:
- Historic Control: The subjects were not enrolled to the control group; data was retrospectively collected by viewing the charts of 20 patients who received Plasma Exchange
Period: Overall Study
Arm/Group | Danazol, Plex, Steroids | Historic Control
Started | 9 | 20
Completed | 8 | 20
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The subjects were not enrolled to the control group; outcome data was retrospectively collected by viewing the charts of 20 patients who received Plasma Exchange. Baseline data was not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Danazol, Plex, Steroids | Historic Control | Total
Number analyzed (Participants) | 9 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.8) |  | 51.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 |  | 3
  Not Hispanic or Latino | 6 |  | 6
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 5 |  | 5
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Plasma Exchanges
Description: The total number of plasma exchanges performed after initiation of the first plasma exchange.
Time Frame: up to 30 days
Measure: Mean (Standard Deviation); unit: exchanges
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 9 | 20
exchanges | 14.8 (9.64) | 16.1 (8.93)

2. Secondary Outcome: Time to Remission
Time Frame: up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 9 | 20
days | 11.4 (5.05) | 11.0 (7.06)

3. Secondary Outcome: Length of Stay
Time Frame: up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 8 | 20
days | 27.3 (17.7) | 24.9 (13.1)

4. Secondary Outcome: Number of Participants With Complete and Continuous Response Rate
Time Frame: At 2 Years
Population: Two of the 20 historical controls did not have data for hospitalization days or time to remission, therefore computed complete response rates among the 18 patients for whom full data was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 9 | 18
Participants
  Complete Response Rate | 9 | 17
  Continuous Response Rate | 8 | 16

5. Secondary Outcome: Time to Relapse
Time Frame: up to 12 years
Measure: Median (Full Range); unit: months
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 1 | 8
months | 43 [NA to NA] — Data for 1 participant, therefore no range | 28.5 [2.5 to 97]

6. Secondary Outcome: Number of Participants With Relapses
Description: Number of participants with relapses
Time Frame: up to 12 years
Measure: Count of Participants; unit: Participants
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 9 | 20
Participants | 1 | 4

7. Secondary Outcome: Number of Relapses
Description: Number of relapses
Time Frame: up to 12 years
Measure: Number; unit: relapses
Arm/Group | Danazol, Plex, Steroids | Historic Control
Number analyzed (Participants) | 1 | 4
relapses | 1 | 6

ADVERSE EVENTS:
Time Frame: 12 years
Description: Adverse events not collected for the historic control arm
Arm/Group | Danazol, Plex, Steroids | Historic Control
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/0
Other Adverse Events (participants affected / at risk) | 0/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danazol, Plex, Steroids (N=9) | Historic Control (N=0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes